CLINICAL TRIAL: NCT04134481
Title: Physiological Responses Related to Clustered Nursing Interventions Among Mechanically Ventilated Patients
Brief Title: Effect Of Clustered Nursing Interventions On Physiological Response In Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Amr Hassan Dahroug, lecturer, critical care medicine, Alexandria University
Other Study IDs: amr dahroug
Record Dates: First submitted 2019-10-16; First posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Mechanically Ventilated Patients
Keywords: clustered nursing interventions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- low intervention group: from 0-7 clustered nursing intervention
- high intervention group: from 8-15 clustered nursing intervention

SUMMARY:
To determine physiological responses related to clustered nursing interventions among critically ill patients.

DETAILED DESCRIPTION:
Clustered nursing interventions are defined as group of interventions more than six for each patient in one nursing interaction.The study was conducted on 80 mechanically ventilated adult patients admitted to intensive care units of Alexandria Main University Hospital and Damanhour Medical National Institute. The most common procedures provided by nurses in direct care for those patients were vital signs measurements, central venous pressure measurement, suctioning, feeding, laboratory sampling, general care, repositioning, and administration of medications. Physiological parameters measured were end-tidal carbon dioxide using capnography, vital signs using bed side monitor, and oxygen saturation using pulse oximeter.

ELIGIBILITY:
Inclusion Criteria:

* adult patients of both sex, aged 18 years and over
* mechanically ventilated for ≥ 48 hours.

Exclusion Criteria:

* lung disorder (eg, COPD, asthma, lung cancer, pneumonia, ARDS)
* pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 80 adult mechanically ventilated patients admitted to intensive care units of Alexandria Main University Hospital (unit I, unit III), General ICU of Damanhur Medical National Institute consists
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2016-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
change in end tidal CO2 in mmHg (EtCO2) change in oxygen saturation (SO2) | up to 14 days
  measured 5 min before procedure (baseline), 5 min after start, 10 min after, immediately at end procedure, 15 min after end procedure for two weeks